CLINICAL TRIAL: NCT01522482
Title: Effects of Meal Fatty Acid Composition on Postprandial Lipaemia in Men According to APOE Genotype
Brief Title: Apolipoprotein (APO)E Genotype, Meal Fatty Acids, Postprandial Lipaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 08/31
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Disease
Keywords: fatty acids; cardiovascular disease; genotype; apoE
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fatty Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High saturated fat meal (Experimental)
  Interventions: Dietary Supplement: High saturated fat meal
- Saturated fatty acid and fish oils meal (Experimental): Equivalent to two portions of oily fish
  Interventions: Dietary Supplement: Saturated fatty acids and fish oil meal
- High unsaturated fat meal (Active Comparator): Provided a fatty acid profile representative of a typical UK diet
  Interventions: Dietary Supplement: High unsaturated fat meal

INTERVENTIONS:
Dietary Supplement: High saturated fat meal — Volunteers consumed a single test meal breakfast containing 53 g of fat, of which 50 g was substituted for saturated fats.
  Arms: High saturated fat meal
Dietary Supplement: Saturated fatty acids and fish oil meal — Volunteers consumed a single test meal breakfast containing 53 g of fat, of which 50 g was substituted for saturated fats and fish oil.
  The dose of fish oils was equivalent to two portions of oily fish.
  Arms: Saturated fatty acid and fish oils meal
Dietary Supplement: High unsaturated fat meal — Volunteers consumed a single test meal breakfast containing 53 g of fat, of which 50 g was substituted for unsaturated fats. It provided a fatty acid profile representative of a typical UK diet.
  Arms: High unsaturated fat meal

SUMMARY:
Cardiovascular disease (CVD) is the greatest cause of morbidity and mortality in the UK. Abnormalities in the concentration and/or composition of lipoproteins (the lipid carrying particles), in particular low density lipoproteins (LDL) in circulation, is one of the most important physiological defects contributing to the development of CVD.

The LDL cholesterol (LDLC) response to fatty acid change is in part mediated by the APOE genotype, with E4 individuals (25% of the UK population) being most responsive to changes in dietary fats, showing greater reductions when low levels of saturated fats or fish oils are consumed and greater increases when high levels of these fats are consumed. Therefore the aims of the present study is to understand the mechanism that regulates the higher LDLC response associated with saturated fatty acids and fish oil consumption in healthy men prospectively recruited based on their APOE genotype.

ELIGIBILITY:
Inclusion Criteria:

* Gender Male
* Age 18-70 years
* Body Mass Index (BMI) < 32 kg/m2
* Plasma triglycerides 1-4 mmol/l
* Plasma cholesterol < 8 mmol/l
* Glucose < 7 mmol/l
* Haemoglobin > 11 g/dl
* ApoE E3/E3, E3/E4

Exclusion Criteria:

* Blood pressure > 200/95 mmHg
* Had suffered a myocardial infraction or stroke in previous 2 years.
* Diabetes mellitus
* Liver disease
* Other endocrine disorders
* Unstable angina
* Familial hyperlipidaemia
* Any dietary restrictions or an a weight reducing diet
* On fatty acid supplements e.g. evening primrose oil or fish oils
* Vigorous exercise e.g. competitive athletes
* ApoE2/E2, apoE2/E3 and apoE2/E4
* Any other parameter on which the investigators felt an individual was unsuitable

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Impact of APOE genotype and dietary fat composition in plasma lipids | 3 months

SECONDARY OUTCOMES:
Cardiovascular disease risk factors | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, Professor, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, United Kingdom

REFERENCES:
- [Derived] Calabuig-Navarro MV, Jackson KG, Kemp CF, Leake DS, Walden CM, Lovegrove JA, Minihane AM. A randomized trial and novel SPR technique identifies altered lipoprotein-LDL receptor binding as a mechanism underlying elevated LDL-cholesterol in APOE4s. Sci Rep. 2017 Mar 9;7:44119. doi: 10.1038/srep44119. PMID 28276521
- [Derived] Calabuig-Navarro MV, Jackson KG, Walden CM, Minihane AM, Lovegrove JA. Apolipoprotein E genotype has a modest impact on the postprandial plasma response to meals of varying fat composition in healthy men in a randomized controlled trial. J Nutr. 2014 Nov;144(11):1775-80. doi: 10.3945/jn.114.197244. Epub 2014 Sep 17. PMID 25332476